CLINICAL TRIAL: NCT03473236
Title: A Phase 1A Single Ascending Dose and Multiple Ascending Dose Double-Blind, Placebo-Controlled, Randomized Trial of Oral Inhalation PK10571 in Healthy Adult Subjects
Brief Title: Phase 1A Safety Trial of Inhaled PK10571 (GB002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GB002, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Collaborators: Pulmokine Inc. (Industry); Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4004002
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Results first posted 2020-02-17 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Safety Issues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (8):
- Cohort 1A (Experimental): Dose 1 Single Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 2A (Experimental): Dose 2 Single Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 3A (Experimental): Dose 3 Single Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 4A (Experimental): Dose 4 Single Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 5A (Experimental): Dose 5 Single Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 1B (Experimental): Dose 1 Multiple Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 2B (Experimental): Dose 2 Multiple Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo
- Cohort 3B (Experimental): Dose 3 Multiple Ascending Dose Protocol: within the cohort, 6 participants receive active drug (GB002) and 2 participants receive placebo.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler; Drug: Placebo

INTERVENTIONS:
Drug: GB002 — Inhaled GB002
  Other Names: PK10571
Device: Generic Dry Powder Inhaler — dry powder inhaler used for inhalation of active drug or placebo
Drug: Placebo — Inhaled placebo

SUMMARY:
This is a phase 1A randomized double blind placebo controlled single ascending dose and multiple ascending dose trial of inhaled PK10571 (GB002) in healthy adult subjects.

DETAILED DESCRIPTION:
This is a first-in-human, single-center, randomized, double-blind, placebo-controlled, two-part study in healthy adult males and females of non-childbearing potential. "Double-Blind" means neither the study subject nor the investigator knows if PK10571 or placebo is being given. "Placebo" means a capsule filled with a powder that does not contain the active drug, PK10571. Because the safety profile of PK10571 in humans is unknown and this is the first clinical study to assess PK10571 in humans, a single-ascending dose design will be used in Part A of the study going from a low dose to higher doses based on safety. Part B will be a multiple-ascending dose design to be run only after review of safety and measurement of drug levels in the blood from Part A.

In the single ascending dose study (Part A) up to five doses may be given to different groups of study subjects based on safety and measurement of drug levels in the blood. Subjects will be randomized into one dose cohort to receive either PK10571 or placebo. Within each cohort, 6 subjects will receive active drug and 2 subjects will receive placebo.

In the multiple ascending dose study (Part B), up to three doses of PK10571 will be tested. The daily dose will be administered daily for 7 days with close clinical monitoring. The dose for the first cohort of Part B will be determined by review of the safety and drug levels from Part A by the Safety Review Committee. The dose interval for the first cohort of Part B (i.e., once daily, twice daily, or up to three times daily) will be determined by review of the safety and drug levels in the blood from Part A by the Safety Review committee. Subsequent doses and dosing intervals will be determined by review of the safety and drug levels from the prior cohort.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (if unable to become pregnant)
* Age 18-55
* Body mass index (BMI) 18-32 kg/m^2 and minimum weight of 50 kg (110 lbs)
* Non-smoker
* Ability to give informed consent
* Ability to remain in study unit for duration of study and return for outpatient visits
* Ability to use dry powder inhaler (DPI) effectively

(See full protocol for additional details.)

Exclusion Criteria:

* Hospitalization within the 6 months prior to the first dose of study treatment
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results
* History or presence of active lung disease (i.e., asthma, chronic obstructive pulmonary disease [COPD], pulmonary fibrosis, hemoptysis, bronchiectasis) or prior intubation
* Currently uses an inhaler
* History or presence of heart disease (i.e., prior myocardial infarction [MI], coronary artery disease, heart failure, hypertension, pulmonary hypertension, valve disease, atrial fibrillation, other arrhythmia, or prolonged QT syndrome)
* History or presence of cancer (with the exception of basal cell skin cancer that has been effectively treated)
* History of diabetes mellitus
* History of thyroid disease other than hypothyroidism control with levothyroxine and documented normal thyroid-stimulating hormone (TSH)
* History of tuberculosis, Lyme disease, or other chronic or opportunistic infection.
* History of positive purified protein derivative (PPD) skin test, or positive PPD test at screening
* Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection
* History of smoking within the past 15 years
* Is a female with a positive pregnancy test result, or who has the ability to become pregnant, or who is lactating
* Has forced expiratory volume in 1 second (FEV1) less than 80% predicted, forced vital capacity (FVC) ˂80% predicted, or resting oxygen saturation less than 97% on room air at screening or baseline
* Upper respiratory infection within the 3 months prior to the first dose of medication
* History of major bleeding or major surgical procedure of any type within 6 months prior to the first dose of medication
* History of minor bleeding disorders such as epistaxis, rectal bleeding (spots of blood on toilet paper), and gingival bleeding within 3 months before the study treatment
* History of bleeding disorder or coagulopathy
* Females with history of dysfunctional uterine bleeding, including history of menorrhagia or metrorrhagia, unless subject has had a hysterectomy.
* History of GI bleed
* Has used any over-the-counter (OTC) medication, nutritional or dietary supplements, herbal preparations, or vitamins within 7 days prior to the first dose of medication
* Has used any antiplatelet agents such as acetylsalicylic acid (ASA), nonsteroidal anti-inflammatory drugs (NSAIDs), clopidogrel (or similar agent) or anti-coagulants within 7 days prior to the first dose of medication
* Has used any prescription medication, except female hormonal replacement therapy, within 14 days prior to the first dose of study medication
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may impact subject safety or the validity of the study results
* History of peripheral vascular disease
* History of autoimmune or collagen vascular disease
* History of sleep apnea
* History of clinically significant allergy to medications
* History of anaphylaxis
* History of liver disease
* History of alcohol or drug abuse
* Prolonged QTc on 12-lead ECG (i.e., QTc corrected using Fridericia's formula [QTcF] ˃450 msec), PR >210 msec, or QRS >110 msec at screening.
* Evidence of prior MI on ECG; presence of atrial fibrillation on ECG; presence of pre-excitation, 2nd or 3rd degree heart block, or abnormal waveform morphology that would preclude accurate measurement of the QT interval duration or other clinically significant abnormalities
* Chest x-ray reveals presence of infiltrate or other abnormality (mass, granuloma, fibrosis, pulmonary thickening, pleural effusion, pulmonary edema, wide mediastinum, cardiomegaly, or clinically significant increased interstitial markings)
* History of neurologic disorder (i.e., multiple sclerosis, amyotrophic lateral sclerosis [ALS], cerebrovascular accident [CVA], transient ischemic attach [TIA])
* History of deep vein thrombosis or pulmonary embolus
* History of clotting disorder
* History of mental illness requiring drug treatment or hospitalization
* History of renal failure or proteinuria (defined as 1+ proteinuria: ≥75 mg/dL on isolated urinalysis)
* Test results greater than the upper limit of normal (ULN) for AST, ALT, or total bilirubin
* Out of range results on the following coagulation tests: INR, prothrombin time (PT), or partial thromboplastin time (PTT)
* Total cholesterol >250 mg/dL or triglycerides >300 mg/dL at screening (based on fasting lipid profile)
* Estimated creatinine clearance less than 60 mL/min
* Hemoglobin at screening of <11.5 g/dl (if female subject) or <12.5 g/dl (if male subject)
* Has a clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening. Note: Subjects with abnormal laboratory results not specifically excluded by this protocol may be enrolled if the Investigator deems the out-of-range values as not clinically significant
* History of treatment with a kinase inhibitor
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication
* Has donated blood or plasma within 30 days prior to the first dose of study medication
* Has participated in another clinical trial (randomized subjects only) within 30 days prior to the first dose of study medication
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine
* Vital signs (measured sitting after 3 minutes rest) at screening that are not within the following ranges (inclusive): heart rate: 40-100 beats per minute [bpm]; systolic blood pressure (BP): 90-145 mmHg; diastolic BP: 50-95 mmHg. Out-of-range vital signs may be repeated once. Blood pressure will be measured in both arms at screening, with a 3-minute rest between each measurement. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing
* Significant difference (i.e., greater than 15 mmHg) between the systolic blood pressure in each arm at screening
* History of lactose intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Phase 1 Unit, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD PK10571 (GB002) Placebo QD: A placebo single ascending dose (SAD) inhaled once a day (QD) over 11 days in healthy volunteers
- SAD GB002 3.75 mg QD: GB002 SAD 3.75 mg inhaled QD over 11 days in healthy volunteers
- SAD GB002 7.5 mg QD: GB002 SAD 7.5 mg inhaled QD over 11 days in healthy volunteers
- SAD GB002 15 mg QD: GB002 SAD 15 mg inhaled QD over 11 days in healthy volunteers
- SAD GB002 30 mg QD: GB002 SAD 30 mg inhaled QD over 11 days in healthy volunteers
- SAD GB002 48 mg QD: GB002 SAD 48 mg inhaled QD over 11 days in healthy volunteers
- MAD GB002 Placebo BID/TID: A placebo multiple ascending dose (MAD) inhaled either twice daily (BID) or thrice daily (TID) over 35 days in healthy volunteers
- MAD GB002 18 mg BID: GB002 MAD 18 mg inhaled BID over 35 days in healthy volunteers
- MAD GB002 24 mg TID: GB002 MAD 24 mg inhaled TID over 35 days in healthy volunteers
- MAD GB002 48 mg TID: GB002 MAD 48 mg inhaled TID over 35 days in healthy volunteers
Period: Overall Study
Arm/Group | SAD PK10571 (GB002) Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Started | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAD GB002 Placebo QD: A placebo SAD inhaled QD over 11 days in healthy volunteers
- MAD GB002 Placebo BID/TID: A placebo MAD inhaled either BID or TID over 35 days in healthy volunteers
- Total: Total of all reporting groups
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (7.72) | 39.0 (7.54) | 36.8 (10.34) | 38.5 (8.78) | 39.5 (6.28) | 35.4 (9.59) | 33.3 (11.31) | 49.3 (4.13) | 31.7 (8.83) | 41.0 (6.10) | 38.8 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 3 | 3 | 32
  Male | 6 | 3 | 3 | 2 | 3 | 4 | 4 | 2 | 4 | 3 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 3 | 4 | 3 | 4 | 4 | 5 | 5 | 3 | 42
  Not Hispanic or Latino | 4 | 1 | 3 | 2 | 3 | 3 | 2 | 1 | 2 | 3 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 1 | 3 | 2 | 0 | 3 | 2 | 2 | 17
  White | 8 | 5 | 5 | 5 | 3 | 5 | 5 | 3 | 5 | 4 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6 | 66
Height [Mean (Standard Deviation); unit: cm] | 172.52 (12.156) | 165.82 (10.699) | 171.03 (14.785) | 169.30 (6.427) | 172.58 (16.351) | 165.84 (11.783) | 169.22 (11.468) | 162.27 (8.190) | 164.43 (9.351) | 167.45 (10.418) | 168.23 (11.220)
Bodyweight [Mean (Standard Deviation); unit: kg] | 79.55 (8.023) | 77.77 (15.075) | 70.37 (16.170) | 76.33 (8.091) | 90.68 (18.925) | 70.37 (6.307) | 81.27 (15.944) | 74.58 (12.449) | 72.24 (8.247) | 65.45 (12.565) | 75.95 (13.255)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.85 (2.804) | 28.07 (3.195) | 23.88 (3.407) | 26.60 (1.932) | 30.18 (1.520) | 25.86 (3.574) | 28.25 (3.384) | 28.18 (2.712) | 26.89 (3.609) | 23.20 (2.589) | 26.79 (3.352)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A serious AE (SAE) is one that, in the view of either the investigator or Sponsor, results in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. A TEAE is defined as any AE that has an onset on or after the first dose of study drug and before the end of study/end of treatment (EoS/ET) visit, or any pre-existing condition that has worsened in severity on or after the first dose of study drug and before the EoS/ET visit.
Time Frame: SAD: from first dose of study drug to 11 days, MAD: from first dose of study drug to 35 days
Population: Safety Population: all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- MAD GB002 Placebo BID/TID: A placebo MAD inhaled either BID or TID to match the dosing in the MAD arms over 35 days in healthy volunteers
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6
Participants
  Any TEAE | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 5 | 4
  Treatment Related TEAE | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 4
  Severe TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious Treatment Related TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE Leading to Early Termination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Vital Sign Findings Reported as TEAEs
Description: Vital signs evaluated included blood pressure, pulse oximetry, respiratory rate, and temperature.
Time Frame: SAD: from first dose of study drug to 11 days, MAD: from first dose of study drug to 35 days
Population: Safety Population: all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Findings in Physical Examinations
Description: Physical examination assessments included: physical exam for general appearance; head, ears, eyes, nose and throat; thyroid; lymph nodes; back and neck; heart; chest; lungs; abdomen; skin; and extremities, musculoskeletal and neurological.
Time Frame: SAD: from first dose of study drug to 11 days, MAD: from first dose of study drug to 35 days
Population: Safety Population: all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in ECG Data (Overall Interpretation)
Description: 12-lead electrocardiograms (ECG) assessments included heart rate, PR interval, QRS duration, QT interval, QTc interval, QTc interval corrected using Bazett's formula (QTcB), QTc interval corrected using Fridericia's formula (QTcF), RR interval.
Time Frame: SAD: Baseline, Day 2, 24 hours; MAD: Baseline, Day 8, 24 hours
Population: Safety Population: all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormal Findings in Pulmonary Function Tests
Description: Pulmonary function tests included forced vital capacity; forced expiratory volume in 1 second (FEV1); forced expiratory flow 25%-75% (FEF25-75); percent predicted forced vital capacity; percent predicted FEV1; and percent predicted FEF25-75.
Time Frame: SAD: from first dose of study drug to 11 days, MAD: from first dose of study drug to 35 days
Population: Safety Population: all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Pharmacokinetic (PK) Analysis of Inhaled GB002: Maximum Concentration (Cmax), SAD
Time Frame: 0 hour (predose), and then at 3, 10, 20, 30, 40 minutes, and 1, 2, 4, 8, 12, 24, 36, and 48 hours after the start of study treatment administration
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 19.4 (41.32) | 51.7 (36.88) | 161 (33.12) | 184 (78.39) | 377 (32.94)

7. Primary Outcome: PK Analysis of Inhaled GB002: Time to Cmax (Tmax), SAD
Time Frame: as for outcome 6
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 0.0833 [0.0833 to 0.0833] | 0.0500 [0.0500 to 0.183] | 0.0500 [0.0500 to 0.0500] | 0.0500 [0.0500 to 0.0500] | 0.0833 [0.0833 to 0.0833]

8. Primary Outcome: PK Analysis of Inhaled GB002: Area Under the Curve From Time 0 Hours to Last Quantifiable Concentration (AUClast), SAD
Time Frame: as for outcome 6
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 28.7 (35.19) | 60.6 (23.01) | 147 (19.51) | 214 (28.55) | 423 (44.51)

9. Primary Outcome: PK Analysis of Inhaled GB002: Area Under the Curve From Time 0 Hours to Infinity (AUCinf), SAD
Time Frame: as for outcome 6
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 28.9 (34.50) | 60.9 (22.90) | 147 (19.43) | 215 (28.48) | 423 (44.41)

10. Primary Outcome: PK Analysis of Inhaled GB002: Apparent Terminal Elimination Half-Life (t1/2), SAD
Time Frame: as for outcome 6
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 3.48 (25.72) | 3.08 (28.54) | 3.32 (12.68) | 4.41 (23.00) | 4.16 (20.35)

11. Primary Outcome: PK Analysis of Inhaled GB002: Apparent Total Plasma Clearance (CL/F), SAD
Description: CL/F is based on nominal (scheduled) dose.
Time Frame: as for outcome 6
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L/h | 130 (34.50) | 123 (22.90) | 102 (19.43) | 140 (28.48) | 113 (44.41)

12. Primary Outcome: PK Analysis of Inhaled GB002: Apparent Volume of Distribution (Vz/F), SAD
Description: Vz/F is based on nominal (scheduled) dose.
Time Frame: as for outcome 6
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L | 650 (25.86) | 548 (24.12) | 489 (18.33) | 889 (32.24) | 681 (44.68)

13. Primary Outcome: PK Analysis of Inhaled GB002: Cmax After Dose 1, MAD
Time Frame: Days 1 and 7: 0 hour (predose), and then at 3, 10, 20, 30, 40 minutes, and 1, 2, 4, 8, 12, 24, 36, and 48 hours after the start of study treatment administration
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 7 | 6
ng/ml
  Day 1 | 146 (35.4) | 229 (55.1) | 571 (26.0)
  Day 7: number analyzed (Participants) | 6 | 6 | 6
  Day 7 | 193 (27.0) | 246 (49.0) | 528 (61.8)

14. Primary Outcome: PK Analysis of Inhaled GB002: Tmax After Dose 1, MAD
Time Frame: as for outcome 13
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 7 | 6
hours
  Day 1 | 0.0833 [0.0833 to 0.0833] | 0.0833 [0.0833 to 0.117] | 0.0833 [0.0833 to 0.0833]
  Day 7: number analyzed (Participants) | 6 | 6 | 6
  Day 7 | 0.0833 [0.0833 to 0.0833] | 0.0833 [0.0833 to 0.0833] | 0.0833 [0.0833 to 0.0833]

15. Primary Outcome: PK Analysis of Inhaled GB002: Area Under the Curve From Time Zero to 24 Hours Postdose (AUC0-24), MAD
Time Frame: as for outcome 13
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 7 | 6
h*ng/mL
  Day 1 | 355 (25.9) | 870 (38.1) | 1690 (39.6)
  Day 7: number analyzed (Participants) | 6 | 6 | 6
  Day 7 | 462 (13.6) | 827 (20.2) | 1870 (42.2)

16. Primary Outcome: PK Analysis of Inhaled GB002: Trough Plasma Concentration (Ctrough), MAD
Time Frame: as for outcome 13
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 7 | 6
h*ng/mL
  Day 1 | 1.27 (65.4) | 2.60 (55.3) | 3.83 (30.4)
  Day 7: number analyzed (Participants) | 6 | 6 | 6
  Day 7 | 2.11 (51.9) | 2.54 (26.0) | 4.29 (24.7)

17. Primary Outcome: PK Analysis of Inhaled GB002: Accumulation Ratio (Rac) for Cmax After Dose 1, MAD
Time Frame: Days 7: 0 hour (predose), and then at 3, 10, 20, 30, 40 minutes, and 1, 2, 4, 8, 12, 24, 36, and 48 hours after the start of study treatment administration
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 6 | 6
ratio | 1.32 (27.3) | 1.13 (24.9) | 0.925 (39.7)

18. Primary Outcome: PK Analysis of Inhaled GB002: Rac for AUC0-24, MAD
Time Frame: as for outcome 17
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 6 | 6
ratio | 1.30 (25.6) | 0.985 (23.5) | 1.11 (16.8)

19. Primary Outcome: PK Analysis of Inhaled GB002: Rac for Ctrough, MAD
Time Frame: as for outcome 17
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 6 | 6
ratio | 1.66 (27.1) | 0.844 (41.0) | 1.12 (19.2)

20. Primary Outcome: PK Analysis of Inhaled GB002: t1/2, MAD
Time Frame: Day 7: 0 hour (predose), and then at 3, 10, 20, 30, 40 minutes, and 1, 2, 4, 8, 12, 24, 36, and 48 hours after the start of study treatment administration
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 6 | 6 | 5
hours | 4.41 (7.04) | 4.68 (18.2) | 5.75 (22.4)

21. Primary Outcome: PK Analysis of Inhaled GB002: Apparent Total Plasma Clearance at Steady-State (CLss/F), MAD
Time Frame: as for outcome 20
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 7 | 7 | 7
L/h | 77.9 (13.55) | 87.1 (20.17) | 76.9 (42.25)

22. Primary Outcome: PK Analysis of Inhaled GB002: Vz/F, MAD
Time Frame: as for outcome 20
Population: PK population: all participants who received active study drug and had at least one quantifiable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 7 | 7 | 7
L | 495 (9.46) | 588 (18.55) | 604 (29.81)

23. Other Pre Specified Outcome: Change From Baseline in White Blood Cell Count
Description: Measurement of white blood cell count
Time Frame: SAD: from baseline to 11 days, MAD: from baseline to 35 days
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
10^9 cells/L | 0.42 (1.212) | -0.07 (1.417) | -0.25 (1.334) | -0.93 (1.694) | -0.75 (1.294) | -0.16 (0.875) | -0.28 (0.768) | 0.27 (0.922) | 0.65 (1.176) | -0.05 (0.689)

24. Other Pre Specified Outcome: Change From Baseline in Hemoglobin
Description: Measurement of hemoglobin
Time Frame: SAD: from baseline to 11 days, MAD: from baseline to 35 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
g/dL | 0.08 (0.573) | -0.62 (0.631) | -0.50 (0.447) | -0.30 (0.721) | 0.00 (0.410) | -0.53 (0.599) | -0.27 (0.683) | -1.13 (0.723) | -1.13 (0.314) | -0.48 (0.512)

25. Other Pre Specified Outcome: Change From Baseline in Kidney Function Parameters
Description: Measurement of blood urea nitrogen (BUN) and creatinine.
Time Frame: SAD: from baseline to 11 days, MAD: from baseline to 35 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
mg/dL
  Change of Urea Nitrogen (BUN) Concentration | -1.50 (3.689) | -0.17 (2.787) | 0.83 (2.994) | -0.17 (2.994) | -0.33 (5.317) | 2.29 (2.289) | 0.00 (4.050) | 0.83 (1.722) | -1.67 (1.966) | -0.33 (3.724)
  Change of Creatinine Concentration | -0.01 (0.099) | 0.03 (0.052) | 0.02 (0.075) | 0.00 (0.089) | 0.03 (0.151) | -0.01 (0.069) | -0.03 (0.052) | -0.07 (0.082) | 0.10 (0.253) | -0.02 (0.041)

26. Other Pre Specified Outcome: Change From Baseline in Liver Function Parameters
Description: Measurement of liver function (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]).
Time Frame: SAD: from baseline to 11 days, MAD: from baseline to 35 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
U/L
  AST | 0.40 (3.098) | -1.17 (5.269) | 2.50 (2.811) | 1.17 (4.750) | 0.17 (2.401) | -1.29 (2.563) | -1.17 (3.125) | -0.67 (3.077) | 1.17 (7.782) | -4.17 (3.430)
  ALT | -0.10 (7.203) | -0.50 (6.025) | 1.17 (1.472) | -0.17 (2.563) | 0.67 (3.204) | -1.14 (4.634) | -2.83 (7.653) | -0.50 (3.886) | 3.50 (13.096) | -2.17 (4.997)

ADVERSE EVENTS:
Time Frame: SAD: from baseline to day 11, MAD: from baseline to day 35
Groups:
- SAD GB002 Placebo QD: A placebo single ascending dose (SAD) inhaled once a day (QD) over 11 days in healthy volunteers
- MAD GB002 Placebo BID/TID: A placebo multiple ascending dose (MAD) inhaled either twice daily (BID) or thrice daily (TID) to match the dosing in the MAD arms over 35 days in healthy volunteers
Arm/Group | SAD GB002 Placebo QD | SAD GB002 3.75 mg QD | SAD GB002 7.5 mg QD | SAD GB002 15 mg QD | SAD GB002 30 mg QD | SAD GB002 48 mg QD | MAD GB002 Placebo BID/TID | MAD GB002 18 mg BID | MAD GB002 24 mg TID | MAD GB002 48 mg TID
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 2/6 | 1/6 | 2/6 | 1/7 | 2/6 | 1/6 | 5/7 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAD GB002 Placebo QD (N=10) | SAD GB002 3.75 mg QD (N=6) | SAD GB002 7.5 mg QD (N=6) | SAD GB002 15 mg QD (N=6) | SAD GB002 30 mg QD (N=6) | SAD GB002 48 mg QD (N=7) | MAD GB002 Placebo BID/TID (N=6) | MAD GB002 18 mg BID (N=6) | MAD GB002 24 mg TID (N=7) | MAD GB002 48 mg TID (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03473236/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03473236/SAP_001.pdf